CLINICAL TRIAL: NCT06823349
Title: Comparative Analysis of Analgesic Efficacy and Maternal Satisfaction: Single Shot Intrathecal Bupivacaine With Fentanyl Versus Bupivacaine With Dexmedetomidine in Normal Labor, Randomized Control Clinical Trial
Brief Title: Comparative Analysis of Analgesic Efficacy: by Single Shot Intrathecal Analgesia (SSSA) in Normal Labor
Acronym: SSSA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jehan George Sadek (Other)
Responsible Party: Sponsor-Investigator, Jehan George Sadek, resident doctor at anesthesia, surgical intensive care unit and pain management department at Aswan University hospital., Aswan University Hospital
Organization: Aswan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Asw.Uni. / 926 / 5 / 24
Record Dates: First submitted 2025-01-20; First posted 2025-02-12 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-01

CONDITIONS: Vaginal Delivery; Normal Labor
Keywords: painless normal labor; Single shot spinal analgesia in vaginal delivery
MeSH Terms: interventions — Dexmedetomidine; Fentanyl; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dexmedetomidine (Active Comparator): the investigators give 5 mic of dexmedetomidine (0.5 ml) added to 2.5 mg bupivacaine (0.5 ml) as total volume 1 ml intrathecally
  Interventions: Drug: Dexmedetomidine
- fentanyl (Active Comparator): the investigators give 25 mic of fentanyl (0.5 ml) added to 2.5 mg bupivacaine (0.5 ml) as total volume 1 ml intrathecally
  Interventions: Drug: fentanyl
- Bupivacaine only (Placebo Comparator): the investigators give 0.5 ml saline 0.9% added to 2.5 mg of bupivacaine (0.5 ml) as total volume 1 ml intrathecally
  Interventions: Drug: Saline 0.9%

INTERVENTIONS:
Drug: Dexmedetomidine — 5 mic dexmedetomidine will be given intrathecally added to 2.5 mg bupivacaine
  Arms: Dexmedetomidine
Drug: fentanyl — 25 mic of fentanyl will be given intrathecally added to 2.5 mg bupivacaine
  Arms: fentanyl
Drug: Saline 0.9% — 0.5 ml of saline 0.9% will be given intrathecally added to 2.5 mg of bupivacaine
  Arms: Bupivacaine only

SUMMARY:
the goal of this randomized control trial is to compare the effect of adding fentanyl v.s dexmedetomidine to bupivacaine in single shot spinal analgesia in achievement of analgesia by decreasing visual analogue scale, onset and increasing duration of analgesia in normal labor.

DETAILED DESCRIPTION:
on arrival to the operating room, the demographic and baseline data will be collected, which include sections about age, height, weight, primigravida or multigravida, cervical dilation at the time of performing labor analgesia, fetus presentation, presence of rupture of membrane, baseline pain scores will be assessed using a 10-cm VAS (0 = no pain and 10 = worst imaginable pain) before SSSA. Intravenous access will be achieved in all patients loading will be undertaken using 500 ml Ringer's solution, baseline values of pulse rate (PR), respiratory rate (RR), hemoglobin oxygen saturation (SpO2), and arterial blood pressure (ABP) will be recorded. SSSA will be performed with the parturient in the sitting position under complete aseptic precautions at the L3-L4 level using a 25-gauge spinal needles. The correct positioning of the needle tip in the intrathecal space will be confirmed by the observation of a free flow of cerebrospinal fluid, and then the prefilled study drug will be injected intrathecally which is 2.5 mg bupivacaine plus 25 mic fentanyl or 5 mic dexmedetomidine or 0.5 ml saline according to different groups.

parturient will then turn to the supine position, and a wedge will be placed under the right buttocks to prevent aortocaval compression. VAS will be evaluated every 5 min for the first 30 min, followed by every 20 min for 3 hours then every 30 min for next 3 hours. If VAS 8 or more the instigators will give the patient 50 mg intramuscular pethidine.

Maternal blood pressure, heart rate, respiratory rate, and oxygen saturation will be measured and recorded noninvasively every 5 min for the first half hour, followed by every 20 min for 3 hours, then every 1 h for next 3 hours. the investigators will give 5 mg ephedrine if there is hypotension ( decrease in ABP more than 25% of the baseline ABP) and .5 mg atropine if there is bradycardia (HR less than 50 beats per minute). Side effects such as hypotension, nausea, vomiting, bradycardia, shivering, pruritus, and tachycardia will be recorded. The first- and fifth-minute Apgar scores will also be recorded. The onset, duration of analgesia, and obstetric and neonatal outcomes will be compared.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II.
* Uncomplicated pregnancy.
* At term & singleton fetus.
* Cervical dilatation > 5cm
* Cephalic presentations

Exclusion Criteria:

* Patient refusal.
* Bleeding disorders and patients on anticoagulant drugs.
* Infection at site of injection.
* Spine deformity.
* Allergy to any of study medications.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
the duration and onset of analgesia. | baseline, pre intervention and after intervention for an average 6 hours
  onset of analgesia will be determined as time taken (in minutes) from the administration of intrathecal drug to the patient reporting effective pain relief (e.g. vas score reduction) duration of analgesia will be determined as time ( in minutes) from onset of analgesia until the patient require additional analgesia or reports significant pain (e.g. VAS score above a threshold).
the change in visual analogue scale (VAS) of the labor pain. | baseline, pre intervention and after intervention an average 6 hours
  change in visual analogue score (VAS) as it is score for measuring pain intensity consisting of 0 to 10 cm line with endpoints labeled as 0 is no pain and 10 is the worst pain and will be evaluated every 5 min for the first 30 min, followed by every 20 min for 3 hours then every 30 min for next 3 hours

SECONDARY OUTCOMES:
maternal satisfaction assessed using a satisfaction questionnaire. | At delivery/birth
  it is a questionnaire that has been made according to 5 scale questionnaire as 1-is very dissatisfied 2- dissatisfied 3- neutral 4- satisfied 5- very satisfied.
change in maternal hemodynamics as blood pressure. | baseline, pre intervention and after intervention for an average 6 hours
  Maternal blood pressure will be measured and recorded noninvasively every 5 minutes for the first half hour, followed by every 20 minutes for 3 hours, then every 1 hour for next 3 hours.
  a hypotension will be defined as ( decrease in mean ABP more than 25% of the baseline mean ABP).
change in maternal hemodynamics as heart rate | baseline, pre intervention and after intervention for an average 6 hours
  heart rate will be measured and recorded noninvasively every 5 minutes for the first half hour, followed by every 20 minutes for 3 hours, then every 1 hour for next 3 hours. a bradycardia will be defined as (HR less than 50 beats per minute).
change in maternal hemodynamics as respiratory rate. | baseline, pre intervention and after intervention for an average 6 hours.
  respiratory rate will be measured and recorded noninvasively every 5 minutes for the first half hour, followed by every 20 minutes for 3 hours, then every 1 hour for next 3 hours. Bradypnea will be defined as respiratory rate below 12 cycle / minute.
Apgar score at 1 and 5 minutes. | will be recorded 1 minute after delivery and 5 minutes after delivery.
  score range 0-10, assessing skin color, heart rate, reflexes, muscle tone, respiratory effort and rate. total score range from 0 to 10. a score of 7 or above indicate good health, while a lower score may require medical attention.

CONTACTS AND LOCATIONS:
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No